CLINICAL TRIAL: NCT02809469
Title: Optimal Dosing of Apixaban in Patients at Risk of Elevated Drug Levels: A Study Evaluating a Strategy of Apixaban Drug Level Measurement and Dose Reduction in Patients With Atrial Fibrillation Who Are at Risk of Elevated Drug Levels
Brief Title: Apixaban Dose Reduction in Patients With Elevated Drug Levels
Acronym: ADREL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ADREL
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose reduction (Experimental): Eligible patients with apixaban levels persistently above 170ng/mL on two occasions, 2 weeks apart, will undergo apixaban dose reduction.
  Interventions: Drug: apixaban dose reduction

INTERVENTIONS:
Drug: apixaban dose reduction — Participants taking apixaban 5mg BID will have their dose reduced to 2.5mg BID, and those taking 2.5mg BID will have their dose reduced to 2.5mg once daily (in the morning).
  Other Names: Eliquis dose reduction

SUMMARY:
Apixaban is an anticoagulant which is increasingly being used to prevent stroke in atrial fibrillation (AF). Phase III clinical trials have demonstrated that apixaban is efficacious and safe for the overall AF population; however, patients older than age 85, with creatinine clearance <40mL/min, or who weighed <50kg were poorly represented in these trials, yet they are commonly seen in real-world clinical scenarios. Advanced age, poor renal function, and low body weight are all associated with elevated drug levels, and elevated drug levels are associated with an increased risk of bleeding. Therefore, clinicians are concerned about the risk of bleeding and are unsure of how best to treat this patient population. Although other anticoagulants are available, apixaban is attractive because it has a low rate of bleeding, low dependence on the kidneys for clearance, and does not require frequent ongoing monitoring and dose adjustment. This study will include patients taking apixaban who were not well-represented in phase III trials - those with age >85, creatinine clearance <40mL/min, or weight <50kg - who are also at increased risk of having elevated drug levels due to these clinical characteristics. Participants will have apixaban levels measured, and those with persistently elevated levels will have their dose reduced. Drug levels will be measured again after dose reduction to determine if the levels are reduced without becoming dangerously low.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular atrial fibrillation (permanent, paroxysmal, or persistent) receiving apixaban with any of the following characteristics: age>85; creatinine clearance <40mL/min; or body weight <50kg.

Exclusion Criteria:

* Inability to visit Hamilton General Hospital;
* Inability or unwillingness to provide written informed consent.
* Stroke or thromboembolic event in the past 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve target range | 1 week after dose reduction
  Patients who undergo dose reduction will have their apixaban drug level measured one week later. The proportion who develop levels between 50-170ng/mL after dose reduction will be determined.

SECONDARY OUTCOMES:
Proportion of patients with persistently elevated levels | 2 weeks after initial blood work
  Patients meeting inclusion criteria will have apixaban drug levels measured. Those with levels above 170ng/mL will have levels repeated 2 weeks later. The proportion of eligible patients with levels above 170ng/mL on both occasions will be determined.
Proportion of patients who spontaneously develop levels below the median of the observed on-therapy range | 2 weeks after initial blood work
  Patients meeting inclusion criteria will have apixaban drug levels measured. Those with levels above 170ng/mL will have levels repeated 2 weeks later. The proportion of patients with levels above 170ng/mL on the first measurement who spontaneously develop levels below 122ng/mL on the second measurement will be determined.
Proportion of patients who develop low levels after dose reduction | 1 week after dose reduction
  Patients who undergo dose reduction will have apixaban drug levels measured 7-10 days after dose reduction. The proportion of patients with drug levels below 50ng/mL after dose reduction will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Vinai C. Bhagirath, MD MSc., Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No